CLINICAL TRIAL: NCT03760263
Title: Evaluation Dose Adjustments in Kidney Transplant Patients on Immediate Release and Extended Release Tacrolimus
Acronym: EVOKE-RT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sentara Norfolk General Hospital (Other)
Collaborators: Veloxis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-19-2018
Record Dates: First submitted 2018-11-03; First posted 2018-11-30 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Transplant;Failure,Kidney
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Envarsus (Active Comparator): Once-daily extended-release tacrolimus
  Interventions: Drug: Tacrolimus
- Prograf (Active Comparator): twice-daily tacrolimus
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Immunosuppressive drug that can prevent organ rejection after transplant in its oral form.
  Other Names: Envarsus

SUMMARY:
Evaluation Dose Adjustments in Kidney Transplant Patients on Immediate Release and Extended Release Tacrolimus

DETAILED DESCRIPTION:
1. Background and Rationale- The novel once-daily extended-release tacrolimus (ERT) has been shown to be non-inferior to twice-daily tacrolimus (TDT) during induction immunotherapy for kidney transplantation. The ERT (Envarsus) has a MeltDose technology that allows for steadier absorption of tacrolimus throughout the entire gastrointestinal tract. This drug has decreased peak to trough fluctuation. This decrease in variability and stabilized trough level should allow for easier achievement of target drug levels with fewer clinic visits and drug level assays.
2. Objective

   1. To assess the safety of ERT versus TDT and effectiveness in achieving tacrolimus trough therapeutic range during the first 6 months after transplantation
   2. Primary End-Point

   i. Ability to achieve center specific target tacrolimus trough levels at the determined intervals after transplantation.

1. Percent of levels in range 2. As most levels occur in the first 6 months, a 6-month time frame will be used for the primary analysis.

c. Secondary End-Points i. Number of dose adjustments required ii. Time in therapeutic range for tacrolimus trough levels during intervals after transplantation based on the Rosendaal Method

1. Time within goal for each time period
2. Time within larger goal of 6-11 iii. Number of lab draws required to achieve trough tacrolimus levels iv. Time to get in therapeutic range v. Cost associated with maintaining therapeutic troughs of tacrolimus
3. Subject Selection a. Subjects will be selected from patients scheduled to receive a living donor or deceased donor kidney transplants at Sentara Norfolk General Hospital b. Inclusion Criteria i. Age 18-70 ii. Receiving a kidney transplant at Sentara Norfolk General Hospital iii. Able to give informed consent c. Exclusion Criteria i. Multi-organ transplant ii. Previous functioning transplant iii. Prior surgery to the gastrointestinal tract that alters the normal anatomy with the exception of cholecystectomy iv. Women of childbearing potential who cannot or are unwilling to maintain adequate contraception during the course of this study.

   d. Patients will be offered enrollment in the study prior to transplant and Informed Consent will be obtained.

   e. Patients will be randomized to standard twice-daily tacrolimus (Prograf) or once-daily extended-release tacrolimus (Envarsus) at a ratio of 1:2.
4. Methods a. Informed Consent to participate in this study will be obtained prior to transplant.

   b. Study subjects will receive usual care induction immunosuppression with Anti-thymocyte globulin or basiliximab, steroids and mycophenolate per the center's protocol.

   c. Subjects enrolled in the study will be randomized and started on tacrolimus within 72 hours after transplant.

   i. Randomization

<!-- -->

1. Prior to study initiation, numbered packets will be created including randomized group and the Informed Consent Form.
2. The packets will be used in order.
3. The group will be determined using the random number generator using values from 1-99 where a value of 1-66 will have an ERT assignment in the study packet and a value of 67-99 will have a TDT assignment in the study packet.

   ii. Subjects randomized to the study group will start ERT at 8mg (or 4mg if concern for delayed graft function) as a single daily dose.

   iii. Subjects randomized to the control group will start TDT at 8mg (or 4mg if concern for delayed graft function) divided in half for a dose every 12 hours.

   iv. If a subject weighs less than or equal to 55kg, then the subject will receive a reduced dose of either ERT or TDT at the provider's discretion.

   d. Subjects' tacrolimus levels in the study will follow our regular post-transplant care. This center uses an outpatient nursing protocol for most patients. If a patient is excluded from the nursing protocol, their tacrolimus levels will be managed individually and changes will be made at the nephrologist's discretion.

   i. Prograf protocol (appendix A) ii. Envarsus protocol (appendix B) e. All other care is routine (nothing done solely for the purpose of research). Other routine care includes: i. Weekly clinic visits and labs for the first month, every other week for the second month then a minimum of monthly through 6 months post transplant.

   ii. During those visits, labs will be drawn, including a tacrolimus level, regardless of study arm. Subjects will receive our routine nephrologist and nurse visits while in clinic. Other specialists (surgeon, dietician, pharmacist, diabetes educator) will see the subjects, as needed.

   iii. Dose changes will either be made in clinic or with a phone call to the subject after clinic, if necessary. Tacrolimus dose changes will be directed by our nurse protocols (appendix A and B). If the subject is excluded from the nursing protocol, the level and dose will be managed by the nephrologist.

5. Investigator Responsibilities- The principal investigator will be responsible to ensure that:

1. all IRB required training for staff and investigators is completed,
2. all staff and investigators comply with the institution's patient and subject safety requirements,
3. the study is conducted in compliance with the protocol and
4. data collection requirements are maintained. 6. Data Analysis

a. Continuous variables will be analyzed using student's t-test or Mann-Whitney U, where appropriate.

b. Categorical variables will be analyzed using the chi2 test or Fischer's Exact test where appropriate.

c. Power analysis for the primary endpoint which will evaluate each level and whether it is in range or not i. Alpha =0.05, beta =0.8 ii. Prior data shows 41% of levels in range for TDT. We predict that ERT dosing will have 53% of levels in range.

iii. With a ratio of 2:1, the minimum will need 406 ERT levels (~38 patients) and 203 TDT levels (~19 patients).

iv. The number of patients is based on patients having 11 levels in the first 6 months, the minimum number of based on our protocol.

7. Data collected includes : i. Inclusion/Exclusion

1. If excluded, reason for exclusion ii. Randomization to Prograf or Envarsus iii. Demographic information

1. Age
2. Height
3. Weight
4. Gender
5. Race
6. Induction (thymoglobulin/basiliximab)
7. CMV donor/recipient exposure status (+/+, +/-, -/+, or -/-)
8. Living or deceased donor iv. Transplant outcomes

1. Rejection (Yes/No and if yes, time interval post-transplant in days). Defined as requiring steroids, thymoglobulin, and/or IVIG 2. BK viremia (Yes/No and if yes, time interval post-transplant in days) 3. CMV viremia (Yes/No and if yes, time interval post-transplant in days) v. Tacrolimus level with time interval post-transplant in days (Yes/No/Not timed correctly) vi. Tacrolimus dose 8. HIPPA Concerns

1. This study will collect data on patient demographics, treatments and outcomes of treatments. Patient data collected will be de-identified of Protected Health Information (PHI) and will not alter patient treatment. This study is designed to address fully HIPAA's requirements for health data that are collected with patient consent.
2. Study data may be made available to third parties, e.g., in the case of an audit performed by regulatory authorities, provided the data are treated confidentially and that the subject's privacy is guaranteed.
3. Subjects identities will not be identifiable or disclosed if results from the study are published.

   9. Data handling

a. The key to patient coding for identification (see Appendix C) and data collection forms will be kept on a password protected computer in a locked office which is only accessible by the investigators and research assistants. To maintain compliance with IRB requirements, the study data will be maintained for the required period of three years. Once the study is completed and data is retained for a minimum of 3 years per the requirements of the IRB, the identifiable data will be destroyed .

10. Human Subjects

1. Due to the nature of the study, there is a potential risk in regards to breach of patient confidentiality. This will be reduced with the collection of the patient's MRN as the identifier, which will then be given a code (see Appendix C), and the storage of this data on a password protected computer in a locked office. The records will be secured for three years according to Federal regulation.
2. Risks

i. There are risks with blood draws that are bruising, swelling at site, and, in rare cases, nerve damage.

ii. Both formulations of tacrolimus (ERT and TDT) are approved for this indication, prevention of rejection after kidney transplant. Expected adverse events have been identified from approval studies. Any serious adverse events will be reported to Veloxis's safety partner, UBC. The study team has the forms to fill out. Any adverse events that require FDA notification will be reported to MedWatch.

c. Benefits i. Subjects who are randomized to receive ERT will receive 6 months-worth of study drug provided by the drug company. After 6 months, the subject's insurance company will be billed for the drug and patients may be responsible for a copayment.

ii. Subjects will not have to pay to participate in the study. iii. Subjects will not be paid to participate in the study. 11. Request for Support

a. The PI requests a 6-month supply of ERT for each subject randomized to the study group.

b. A request for funding for direct study activities will be requested when the research center and the sponsor have agreed to the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* Receiving a kidney transplant at Sentara Norfolk General Hospital
* Able to give informed consent

Exclusion Criteria:

* Multi-organ transplant
* Previous functioning transplant
* Prior surgery to the gastrointestinal tract that alters the normal anatomy with the exception of cholecystectomy
* Women of childbearing potential who cannot or are unwilling to maintain adequate contraception during the course of this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
I. Percentage of tacrolimus levels in range after transplantation | 6 Months
  Labs will be drawn at weekly clinic visits for the first month, every other week for the second month, then a minimum of monthly through 6 months post transplant. Labs drawn will include tacrolimus level to determine if trough levels are within target ranges according to the site's center specific tacrolimus protocol.

SECONDARY OUTCOMES:
II. Time in therapeutic range for tacrolimus trough levels during intervals after transplantation based on the Rosendaal Method | 6 Months
  Therapeutic range is defined by the site's center specific tacrolimus protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas McCune, MD, Principal Investigator — Sentara Norfolk General Hospital
Locations (1):
- Sentara Norfolk General Hospital, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided